CLINICAL TRIAL: NCT02546167
Title: Pilot Study Of Redirected Autologous T Cells Engineered To Contain an Anti-BCMA scFv Coupled To TCRζ And 4-1BB Signaling Domains in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: CART-BCMA Cells for Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 14415, 822756
Record Dates: First submitted 2015-09-09; First posted 2015-09-10 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): will receive 1-5x10^7 CART-BCMA cells given as a split dose infusion over 3 days.
  Interventions: Biological: CART-BCMA
- Cohort 2 (Experimental): Cyclophosphamide infusion prior to 1-5x10^7 CART BCMA cells given as a split dose infusion over 3 days.
  Interventions: Biological: CART-BCMA
- Cohort 3 (Experimental): Cyclophosphamide infusion prior to 1-5x10^8 CART BCMA cells given as a split dose infusion over 3 days.
  Interventions: Biological: CART-BCMA

INTERVENTIONS:
Biological: CART-BCMA

SUMMARY:
Open-label, single-center, pilot study to assess the safety and feasibility of infusion of autologous T cells expressing BCMA (B-cell maturation antigen)-specific chimeric antigen receptors with tandem TCR and 4-1BB costimulatory domains (referred to as CART-BCMA ) in adult patients with multiple myeloma (MM). CART-BCMA cells will be given as a split dose intravenous infusion over 3 days. The duration of active intervention and monitoring is approximately 2 years.

DETAILED DESCRIPTION:
At entry subjects will undergo routine laboratory and imaging assessment of their multiple myeloma. Eligible subjects will undergo steady-state apheresis to obtain large numbers of peripheral blood mononuclear cells (PBMC) for CART-BCMA manufacturing. Cryopreserved historical apheresis products collected from the patient prior to study entry are usable for CART-BCMA manufacturing if collected at an appropriately certified apheresis center and the product meets adequate mononuclear cell yields. If a historical apheresis product is not available, an apheresis procedure will be scheduled for cell procurement after study entry. The T cells will be purified from the PBMC, transduced with TCRζ/4-1BB lentiviral vector, expanded in vitro and then frozen for future administration. The number of subjects who have inadequate T cell collections, expansion or manufacturing compared to the number of subjects who have CAR T cells successfully manufactured will be recorded; feasibility of product manufacturing is not expected to be problematic in this patient population.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must have a confirmed prior diagnosis of active MM as defined by the updated IMWG criteria101..
2. Subjects must have relapsed or refractory disease after either one of the following:

   1. At least 3 prior regimens, which must have contained an alkylating agent, proteasome inhibitor, and immunomodulatory agent (IMiD).

      OR
   2. At least 2 prior regimens if "double-refractory" to a proteasome inhibitor and IMiD, defined as progression on or within 60 days of treatment with these agents.

   Note: Induction therapy, stem cell transplant, and maintenance therapy, if given sequentially without intervening progression, should be considered as 1 "regimen".
3. Subjects must have signed written, informed consent.
4. Subjects must be ≥ 18 years of age.
5. Subjects must be at least 90 days since autologous or allogeneic stem cell transplant, if performed.
6. Subjects must have adequate vital organ function:

   1. Serum creatinine ≤ 2.5 or estimated creatinine clearance ≥30 ml/min and not dialysis-dependent.
   2. Absolute neutrophil count ≥1000/μl and platelet count ≥50,000/μl (≥30,000/μl if bone marrow plasma cells are ≥50% of cellularity).
   3. SGOT ≤ 3x the upper limit of normal and total bilirubin ≤ 2.0 mg/dl (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome).
   4. Left ventricular ejection fraction (LVEF) ≥ 45%. LVEF assessment must have been performed within 8 weeks of enrollment.
   5. Toxicities from prior therapies, with the exception of peripheral neuropathy attributable to bortezomib, must have recovered to grade ≤ 2 according to the CTC 4.0 criteria or to the subject's prior baseline.
7. Subjects must have an ECOG performance status of 0-2.
8. Subjects must have measurable disease on study entry, which must include at least 1 of the following:

   1. Serum M-spike ≥ 0.5 g/dL*
   2. 24 hr urine M-spike ≥ 200mg
   3. Involved serum FLC ≥ 50 mg/L with abnormal ratio
   4. Measurable plasmacytoma on exam or imaging
   5. Bone marrow plasma cells ≥ 20% (bone marrow biopsy only required at screening if no other measurable disease is present).

      * Note: Patients with IgA myeloma in whom serum protein electrophoresis is deemed unreliable, due to co-migration of normal serum proteins with the paraprotein in the beta region, may be considered eligible as long as total serum IgA level is elevated above normal range.
9. Subjects of reproductive potential must agree to use acceptable birth control methods.

IMWG Criteria for Diagnosis of Multiple Myeloma Presence of an M-component in serum and/or urine plus clonal plasma cells in the bone marrow and/or a documented clonal plasmacytoma. In patients with no detectable M-component, an abnormal serum FLC ratio on the serum FLC assay can substitute and satisfy this criterion. For patients, with no serum or urine M-component and normal serum FLC ratio, the baseline bone marrow must have ≥10% clonal plasma cells; these patients are referred to as having 'non-secretory myeloma'. Patients with biopsy-proven amyloidosis and/or systemic light chain deposition disease (LCDD) should be classified as 'myeloma with documented amyloidosis' or 'myeloma with documented LCDD,' respectively if they have ≥30% plasma cells and/or myeloma-related bone disease.

PLUS one or more of the following, which must be attributable to the underlying plasma cell disorder:

* Calcium elevation (>11.5 mg/dl)
* Renal insufficiency (creatinine >2 mg/dl)
* Anemia (hemoglobin <10 g/dl or at 2 g/dl below normal)
* Bone disease (lytic lesions or osteopenia) OR one of the following "myeloma-defining events"
* Bone marrow plasma cells ≥60% of cellularity
* Serum free kappa:lambda ratio ≥100:1 (or ≤1:100), with involved free light chain ≥100 mg/L
* More than 1 focal bone lesion on MRI

Exclusion Criteria

* Be pregnant or lactating.
* Have inadequate venous access for or contraindications to leukapheresis.
* Have any active and uncontrolled infection.
* Have active hepatitis B, hepatitis C, or HIV infection.
* Any uncontrolled medical or psychiatric disorder that would preclude participation as outlined.
* Have NYHA Class III or IV heart failure, unstable angina, or a history of recent (within 6 months) myocardial infarction or sustained (>30 seconds) ventricular tachyarrhythmias.
* Have received prior gene therapy or gene-modified cellular immunotherapy. Subject may have received, however, non-gene-modified autologous T-cells in association with an anti-myeloma vaccine (e.g., hTERT or MAGEA3) or vaccination against infectious agents (e.g., influenza or pneumococcus) as was performed on our previous studies.
* Have active auto-immune disease, including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the principal investigator) autoimmune disease requiring prolonged immunosuppressive therapy.
* Have a history of neurodegenerative or central nervous system movement disorder.
* Have prior or active central nervous system (CNS) involvement (e.g. leptomeningeal disease, parenchymal masses) with myeloma. Screening for this (e.g. with lumbar puncture) is not required unless suspicious symptoms or radiographic findings are present. Subjects with calvarial disease that extends intracranially and involves the dura will be excluded, even if CSF is negative for myeloma.
* Have active acute or chronic graft-versus-host-disease (GVHD), or require immunosuppressant medications for GVHD, within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-03; Primary Completion 2019-08-21 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years
  Study related adverse events (defined as ≥ Grade 3 signs/symptoms according to CTCAE 4.03, laboratory toxicities, and clinical events) that are "possibly", "probably", or "definitely" related to study treatment any time from the first day of study treatment until end of study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Cohen AD, Garfall AL, Stadtmauer EA, Melenhorst JJ, Lacey SF, Lancaster E, Vogl DT, Weiss BM, Dengel K, Nelson A, Plesa G, Chen F, Davis MM, Hwang WT, Young RM, Brogdon JL, Isaacs R, Pruteanu-Malinici I, Siegel DL, Levine BL, June CH, Milone MC. B cell maturation antigen-specific CAR T cells are clinically active in multiple myeloma. J Clin Invest. 2019 Mar 21;129(6):2210-2221. doi: 10.1172/JCI126397. PMID 30896447
- [Derived] Bu DX, Singh R, Choi EE, Ruella M, Nunez-Cruz S, Mansfield KG, Bennett P, Barton N, Wu Q, Zhang J, Wang Y, Wei L, Cogan S, Ezell T, Joshi S, Latimer KJ, Granda B, Tschantz WR, Young RM, Huet HA, Richardson CJ, Milone MC. Pre-clinical validation of B cell maturation antigen (BCMA) as a target for T cell immunotherapy of multiple myeloma. Oncotarget. 2018 May 25;9(40):25764-25780. doi: 10.18632/oncotarget.25359. eCollection 2018 May 25. PMID 29899820